CLINICAL TRIAL: NCT04307407
Title: The Cause Trial: A Randomized Trial of Aerobic Exercise on CVD Risk Factors in Breast Cancer Survivors
Brief Title: Exercise in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Oslo University Hospital (Other); Memorial Sloan Kettering Cancer Center (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Tormod Skogstad Nilsen, PhD, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/1318
Record Dates: First submitted 2020-03-06; First posted 2020-03-13 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental): The aim is for participants to complete three weekly sessions of supervised aerobic treadmill based exercise for five months. Session duration varies from 20-60 minutes, with exercise intensity ranging from 55-95% of peak heart rate. Maximal exercise capacity (VO2peak and peak heart rate), will be determined by the CPET performed by certified exercise physiologists at baseline.
  Interventions: Behavioral: Aerobic Exercise
- Standard care (No Intervention): Participants in this arm will not receive any follow-up on exercise during the intervention period.
- Reference Group (Other): Participants in this arm are age-matched women with no history of any malignant disease, which will undergo similar assessments at baseline and post-intervention and also follow similar exercise intervention as the breast cancer survivors randomized to the Aerobic exercise arm
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will be randomized to supervised aerobic exercise or standard care. Women with no current or past malignant disease will comprise the reference group and will be matched for age to participants in the Aerobic Exercise arm
  Arms: Aerobic Exercise; Reference Group

SUMMARY:
The purpose of this study is to compare the effects of aerobic exercise to usual care in women treated with chemotherapy and radiation therapy for non-metastatic breast cancer

DETAILED DESCRIPTION:
In this study, we will compare the effects of exercise between women previously treated with breast cancer to women with no history of any cancers. Therefore, in addition to a randomized controlled trial in women with previous breast cancer (i.e., an exerciser group and a control group), we also include a reference group comprising age-matched women with no history of any cancer diagnosis. Women in the reference group will undergo a similar exercise intervention and the exercise group. This study recruits through invitation only.

The primary endpoint in this study is the change in cardiorespiratory fitness, measured as VO2peak. Secondary endpoints include common risk factors for cardiovascular disease and cardiometabolic health, endpoints derived from the cardiopulmonary exercise test and lung function assessments, cellular muscle endpoints derived from muscle biopsies obtained from m. vastus lateralis, also patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible BCS must be listed in the Norwegian Cancer registry
* Female
* Adult-onset breast cancer diagnosis, diagnosed between 2008 and 2012
* 60 years or younger at the time of diagnosis
* received anthracycline-based chemotherapy as a part of their treatment history
* signed informed consent and medical doctors approveal of participation prior to inclusion

Exclusion Criteria:

* Received Herceptin
* Diagnosed with stage IV breast cancer
* Relapse since diagnosis
* A history, or current presence, of another diagnosis of invasive cancer of any kind
* Selfreported severe fatigue
* present with any uncontrolled- or recent cardiovascular disease, has undergone heart surgery or uses a pacemaker
* currently exercising more than 90 minutes per week

Ages: 28 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak | From baseline to five months (post-intervention)
  Peak oxygen uptake during a treadmill based cardiopulmonary exercise test

SECONDARY OUTCOMES:
Systolic- and diastolic heart chamber dimensions | From baseline to five months (post-intervention)
  Cardiac morphology and function will be assessed by 2D and 3D Echocardiography and 2D strain echocardiography
Systolic- and diastolic longitudinal strain | From baseline to five months (post-intervention)
  Cardiac morphology and function will be assessed by 2D and 3D Echocardiography and 2D strain echocardiography
Lean body mass | From baseline to five months (post-intervention)
  Body composition will be assessed by dual x-ray absorptiometry
Fat mass | From baseline to five months (post-intervention)
  Body composition will be assessed by dual x-ray absorptiometry
Blood volume | From baseline to five months (post-intervention)
  Hemoglobin mass and blood volume will be assessed using the carbon monoxide rebreathing method
Muscle fiber type | From baseline to five months (post-intervention)
  Change in muscle morphology will be assessed in muscle biopsies using immunohistochemistry
Muscle fiber area | From baseline to five months (post-intervention)
  Change in muscle morphology will be assessed in muscle biopsies using immunohistochemistry
Muscle mitochondria mass | From baseline to five months (post-intervention)
  Change in mitochondrial proteins will be assessed in muscle biopsies using western blot
Quality of life: Quality of Life Questionnaire (QLQ) C-30 | From baseline to five months (post-intervention)
  Relevant patient reported outcomes will be obtained using validated Quality of Life Questionnaire (QLQ) C-30
Genome-wide DNA methylation and gene expression | From baseline to five months (post-intervention)
  For a sub-group of participants, muscle biopsies will be further processed for RNA and DNA

CONTACTS AND LOCATIONS:
Overall Officials: Tormod S Nilsen, PhD, Principal Investigator — The Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansen SH, Reinertsen KV, Wisloff T, Saeter M, Sarvari SI, Kiserud CE, Strandos N, Edvardsen E, Grydeland M, Nilsen TS, Thorsen L. Effects of aerobic exercise on late effects and quality of life in long-term breast cancer survivors: a randomized controlled trial. JNCI Cancer Spectr. 2025 Nov 3;9(6):pkaf102. doi: 10.1093/jncics/pkaf102. PMID 41117797
- [Derived] Saeter M, Johansen SH, Reinertsen KV, Thorsen L, Haugaa KH, Nilsen TS, Sarvari SI. Cardiorespiratory fitness, cardiac morphology and function, and cardiovascular risk factors in long-term breast cancer survivors compared with non-cancer controls. Cardiooncology. 2025 Jan 4;11(1):1. doi: 10.1186/s40959-024-00296-0. PMID 39755716
- [Derived] Nilsen TS, Saeter M, Sarvari SI, Reinertsen KV, Johansen SH, Edvardsen ER, Hallen J, Edvardsen E, Grydeland M, Kiserud CE, Lie HC, Solberg PA, Wisloff T, Sharples AP, Raastad T, Haugaa KH, Thorsen L. Effects of Aerobic Exercise on Cardiorespiratory Fitness, Cardiovascular Risk Factors, and Patient-Reported Outcomes in Long-Term Breast Cancer Survivors: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 15;12:e45244. doi: 10.2196/45244. PMID 36920460